CLINICAL TRIAL: NCT07094165
Title: Evaluation of the Effects of Remifentanil and Dexmedetomidine on Crush Injury and Renal Functions in an Experimental Model
Brief Title: The Effects of Dexmedetomidine and Remifentanil on Kidney Injury After Muscle Compression Injury in Rats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: AnkaraCHBilkent0741
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury; Crush Injury; Rhabdomyolysis
Keywords: remifentanil; dexmedetomidine; crush injury; renal injury; KIM-1; NGAL
MeSH Terms: conditions — Acute Kidney Injury; Crush Injuries; Rhabdomyolysis | interventions — Dexmedetomidine; Remifentanil; Laparotomy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): The control group did not receive any intervention or pharmacological treatment.
- Dexmedetomidine (Experimental): Following 2 hours of bilateral muscle compression, rats in the dexmedetomidine group underwent a 1-hour period including both laparotomy and continuous intravenous dexmedetomidine infusion.
  Interventions: Drug: Dexmedetomidine; Procedure: Laparotomy; Procedure: Compression
- Remifentanil (Experimental): Following 2 hours of bilateral muscle compression, rats in the remifentanil group underwent a 1-hour period including both laparotomy and continuous intravenous remifentanil infusion.
  Interventions: Drug: Remifentanil; Procedure: Laparotomy; Procedure: Compression
- Sham (Sham Comparator): In the sham group, bilateral gastrocnemius muscle compression was applied for 2 hours and laparotomy was performed, but no pharmacological intervention was given.
  Interventions: Procedure: Laparotomy; Procedure: Compression

INTERVENTIONS:
Drug: Dexmedetomidine — Following 2 hours of bilateral muscle compression, rats in the dexmedetomidine group underwent a 1-hour period including both laparotomy and continuous intravenous dexmedetomidine infusion.
  Arms: Dexmedetomidine
Drug: Remifentanil — Following 2 hours of bilateral muscle compression, rats in the remifentanil group underwent a 1-hour period including both laparotomy and continuous intravenous remifentanil infusion.
  Arms: Remifentanil
Procedure: Laparotomy — A standardized laparotomy was carried out for 1 hour, during which the abdominal cavity was opened and subsequently closed. This procedure aimed to mimic the physiological impact of a one-hour surgical operation.
  Arms: Dexmedetomidine; Remifentanil; Sham
Procedure: Compression — Bilateral compression was applied to the gastrocnemius muscles for a duration of 2 hours.
  Arms: Dexmedetomidine; Remifentanil; Sham

SUMMARY:
The goal of this interventional preclinical study is to evaluate the potential protective effects of two intravenous anesthetic agents-dexmedetomidine and remifentanil-on kidney function in the context of muscle crush injury, which is known to be a major contributor to acute kidney injury (AKI) following trauma, entrapment, or disasters such as earthquakes. AKI following crush syndrome results from rhabdomyolysis, hypovolemia, oxidative stress, and systemic inflammation, and it significantly increases morbidity and mortality. This study explores whether anesthetic choice during the acute phase of injury influences renal outcomes.

This study used a rat model of crush injury. A total of 28 healthy adult male Wistar rats were randomly divided into four groups (n=7 per group):

1. Control group - no surgical procedure, no injury, no drug.
2. Sham group - anesthesia and cannulation were performed but no crush injury or drug administered.
3. Dexmedetomidine group - crush injury + intravenous dexmedetomidine infusion (3 µg/kg/h) for 1 hour.
4. Remifentanil group - crush injury + intravenous remifentanil infusion (1 µg/kg/h) for 1 hour.

Crush injury was induced by applying a metal clamp with a constant pressure of 3 kg to both gastrocnemius muscles for 2 hours, under anesthesia. After the clamp was removed, animals in the two treatment groups received a one-hour intravenous infusion of their assigned drug. Blood samples were taken at baseline and at 6 hours post-injury. After euthanasia, bilateral kidney tissues were harvested for biochemical and histopathological evaluation.

The main questions this study aimed to answer were:

* Does dexmedetomidine reduce serum and tissue levels of AKI biomarkers (such as NGAL, KIM-1, TIMP-2, IGFBP7) more effectively than remifentanil in a rat model of crush injury?
* Are there histological differences in kidney damage between the treatment groups?
* What is the impact of both drugs on oxidative stress markers (TAC - total antioxidant capacity, TOS - total oxidant status) and renal function parameters such as creatinine and urea?

Biochemical analyses included ELISA-based quantification of NGAL, KIM-1, TIMP-2, IGFBP7, TAC, TOS, serum creatinine, and BUN. Histopathological scoring was performed by a blinded pathologist, assessing tubular necrosis, interstitial edema, and inflammatory cell infiltration.

The study found that rats in the dexmedetomidine group exhibited lower levels of renal injury markers and histopathological damage scores compared to those in the remifentanil group. These findings suggest that dexmedetomidine may offer superior renal protection during acute crush injury compared to remifentanil, potentially via anti-inflammatory and antioxidant mechanisms.

The results of this study may help guide anesthetic drug selection in trauma patients at high risk of kidney injury, and lay the foundation for future translational research.

ELIGIBILITY:
Rat Experiment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Serum Creatinine Level | Baseline (0 hour), 2 hours, and 6 hours after intervention
  Change in serum creatinine levels measured at 0, 2, and 6 hours after experimental crush injury in Wistar Albino rats receiving either dexmedetomidine or remifentanil. This outcome is used to assess renal function and the nephroprotective effect of the interventions.

SECONDARY OUTCOMES:
Neutrophil Gelatinase-Associated Lipocalin (NGAL) Level | 0, 2, and 6 hours after intervention
  NGAL levels measured in serum at three time points to assess early renal tubular injury following experimental crush injury and treatment with dexmedetomidine or remifentanil. NGAL is an early biomarker for acute kidney injury (AKI) and reflects renal stress.
Histopathological Tubular Injury Score | At 6 hours after intervention (after sacrifice)
  Histopathological evaluation of renal tissue samples using scoring for tubular necrosis, brush border loss, dilatation, congestion, and apoptotic cell count. Quantitative damage scoring was performed blindly by two pathologists to compare the nephroprotective effects of dexmedetomidine and remifentanil.
Kidney Injury Molecule-1 (KIM-1) Level | 0, 2, and 6 hours after intervention
  Serum levels of KIM-1 measured by ELISA to evaluate renal tubular epithelial injury and compare the protective effects of the two anesthetic agents.
TIMP-2) × (IGFBP7) Product Level | The combined serum levels of TIMP-2 and IGFBP7, representing G1 cell cycle arrest, were measured to detect early renal stress and predict AKI development in the experimental model.
  0, 2, and 6 hours after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a preclinical animal study conducted on Wistar Albino rats. Since no human subjects were enrolled, there is no individual participant data (IPD) to share.

REFERENCES:
- [Result] Bao N, Dai D. Dexmedetomidine Protects against Ischemia and Reperfusion-Induced Kidney Injury in Rats. Mediators Inflamm. 2020 Apr 3;2020:2120971. doi: 10.1155/2020/2120971. eCollection 2020. PMID 32317860
- [Result] Bywaters EG, Beall D. Crush Injuries with Impairment of Renal Function. Br Med J. 1941 Mar 22;1(4185):427-32. doi: 10.1136/bmj.1.4185.427. No abstract available. PMID 20783577
- [Result] Bostankolu E, Ayoglu H, Yurtlu S, Okyay RD, Erdogan G, Deniz Y, Hanci V, Can M, Turan IO. Dexmedetomidine did not reduce the effects of tourniquet-induced ischemia-reperfusion injury during general anesthesia. Kaohsiung J Med Sci. 2013 Feb;29(2):75-81. doi: 10.1016/j.kjms.2012.08.013. Epub 2012 Oct 13. PMID 23347808
- [Result] Celikmen MF, Sarikaya S, Ozucelik DN, Sever MS, Aciksari K, Celikmen DM, Yazicioglu M, Kandemir A, Dogan H, Ayvaci BM, Ozasir Abuska D, Sadillioglu S. Effects of acetaminophen and mannitol on crush injuries in rats: An experimental study. Ulus Travma Acil Cerrahi Derg. 2016 Jul;22(4):305-14. doi: 10.5505/tjtes.2015.76824. PMID 27598600
- [Result] de Carvalho AL, Vital RB, Kakuda CM, Braz JR, Castiglia YM, Braz LG, Modolo MP, Ribeiro OR, Domingues MA, Modolo NS. Dexmedetomidine on renal ischemia-reperfusion injury in rats: assessment by means of NGAL and histology. Ren Fail. 2015 Apr;37(3):526-30. doi: 10.3109/0886022X.2015.1006118. Epub 2015 Jan 23. PMID 25613736
- [Result] Erkilic E, Kesimci E, Alaybeyoglu F, Kilinc I, Tural R, Yazgan A, Gumus T, Sepici Dincel A, Dumlu EG, Kanbak O. Does remifentanil attenuate renal ischemia-reperfusion injury better than dexmedetomidine in rat kidney? Drug Des Devel Ther. 2017 Mar 8;11:677-683. doi: 10.2147/DDDT.S126701. eCollection 2017. PMID 28331287
- [Result] Gonullu E, Ozkardesler S, Kume T, Duru LS, Akan M, Guneli ME, Ergur BU, Meseri R, Dora O. Comparison of the effects of dexmedetomidine administered at two different times on renal ischemia/reperfusion injury in rats. Braz J Anesthesiol. 2014 May-Jun;64(3):152-8. doi: 10.1016/j.bjane.2013.06.002. Epub 2013 Oct 16. PMID 24907872
- [Result] Kanbak O, Aydogan B, Gumus T. Effects of remifentanil and propofol on distant organ lung injury in an ischemia-reperfusion model. Open Med (Wars). 2021 Nov 8;16(1):1673-1680. doi: 10.1515/med-2021-0381. eCollection 2021. PMID 34761118
- [Result] Kocoglu H, Ozturk H, Ozturk H, Yilmaz F, Gulcu N. Effect of dexmedetomidine on ischemia-reperfusion injury in rat kidney: a histopathologic study. Ren Fail. 2009;31(1):70-4. doi: 10.1080/08860220802546487. PMID 19142813
- [Result] Sugita S, Okabe T, Sakamoto A. Continuous infusion of dexmedetomidine improves renal ischemia-reperfusion injury in rat kidney. J Nippon Med Sch. 2013;80(2):131-9. doi: 10.1272/jnms.80.131. PMID 23657066
- [Result] Si YN, Bao HG, Xu L, Wang XL, Shen Y, Wang JS, Yang XB. Dexmedetomidine protects against ischemia/reperfusion injury in rat kidney. Eur Rev Med Pharmacol Sci. 2014 Jul;18(13):1843-51. PMID 25010612

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT07094165/Prot_SAP_000.pdf